CLINICAL TRIAL: NCT02607813
Title: A Phase I Dose Finding Study of Oral LXH254 in Adult Patients With Advanced Solid Tumors Harboring MAPK Pathway Alterations
Brief Title: Phase I Study of LXH254 in Patients With Advanced Solid Tumors Haboring MAPK Pathway Alterations
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLXH254X2101; 2015-003421-33 (EudraCT Number)
Record Dates: First submitted 2015-11-05; First posted 2015-11-18 (Estimated); Last update posted 2022-12-21 (Actual); Status verified 2022-03

CONDITIONS: NSCLC; Ovarian Cancer; Melanoma; Other Solid Tumors
Keywords: LXH254, CRAF, MAPK, solid tumor, PDR001
MeSH Terms: conditions — Ovarian Neoplasms; Melanoma | interventions — naporafenib; spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Dose escalation LXH254 (Experimental)
  Interventions: Drug: LXH254
- Dose expansion LXH254: Group 1 (Experimental)
  Interventions: Drug: LXH254
- Dose expansion LXH254: Group 2 (Experimental)
  Interventions: Drug: LXH254
- Dose expansion LXH254: Group 3 (Experimental)
  Interventions: Drug: LXH254
- Dose expansion: LXH254 + PDR001 (Experimental)
  Interventions: Drug: LXH254; Drug: PDR001
- Dose escalation LXH254 + PDR001 (Experimental)
  Interventions: Drug: LXH254; Drug: PDR001

INTERVENTIONS:
Drug: LXH254 — pan-RAF inhibitor
Drug: PDR001 — Biological: PDR001 anti-PD1 antibody
  Arms: Dose escalation LXH254 + PDR001; Dose expansion: LXH254 + PDR001

SUMMARY:
A Phase I Study of LXH254 in Patients With Advanced Solid Tumors That Harbor MAPK Pathway Alterations.

ELIGIBILITY:
Inclusion Criteria:

* All patients participating in this clinical trial must have progressed following standard therapy, or for whom, in the opinion of the Investigator, no effective standard therapy exists, is tolerated or appropriate.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
* Presence of at least one measurable lesion according to RECIST v1.1.
* Documented MAPK alteration

Additional inclusion criteria for the Dose Expansion part: LXH254 in combination with PDR001:

* Patients with confirmed KRAS-mutated NSCLC
* Patients with confirmed NRAS-mutated melanoma (cutaneous melanoma only)

Exclusion Criteria:

- Prior treatment with a BRAFi, MEKi and/or pan-RAF inihibitors for patients to be enrolled in the dose expansion part.

Exceptions may be made after documented agreement between Novartis and Investigator.

* History or current evidence of retinal vein occlusion (RVO) or current risk factors for RVO.
* Any medical condition that would, in the investigator's judgment, prevent the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures.
* Patients receiving proton pump inhibitors which cannot be discontinued 3 days prior to the start study treatment and for the duration of the study.
* Pregnant or nursing (lactating) women

Additional exclusion criteria for LXH254 in combination with PDR001

* History of severe hypersensitivity reactions, which in the opinion of the investigator may cause in increased risk of serious infusion reaction.
* Known human immunodeficiency virus (HIV).
* Any positive test for hepatitis B virus or hepatitis C virus indicating acute or chronic infection.
* Active, known or suspected autoimmune disease.
* Active infection requiring systemic antibiotic therapy
* Patients requiring systemic steroid therapy or any immunosuppressive therapy (≥10mg/day prednisone or equivalent) which cannot be discontinued at least 7 days prior to first dose of study treatment.
* Use of any live vaccines against infectious diseases within 4 weeks of initiation of study treatment.

Other inclusion/exclusion criteria as per protocol may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2016-01-18 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-02-19 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability as assessed by incidence and severity of adverse events (AEs), dose interruptions, reductions, and dose intensity. | From Cycle 1 Day 1 until 30 days for LXH254 single agent and 150 days for LXH254 in combination with PDR001 post study treatment (expected duration approximately 12 months)
  cycle = 28 days
Incidence and nature of dose limiting toxicities (DLTs) (dose escalation and LXH254 single agent only) | 28 days
  cycle = 28 days
Incidence and nature of dose limiting toxicities (DLTs) (dose escalation and LXH254 in combination with PDR001 only) | 56 days
  cycle =28 days

SECONDARY OUTCOMES:
Overall response rate (ORR) | Every 2 cycles after starting study treatment until end of treatment; expected duration approximately 12 months
  cycle = 28 days
Disease control rate (DCR) | Every 2 cycles after starting study treatment until end of treatment; expected duration approximately 12 months
  cycle = 28 days
Duration of response (DoR) | Every 2 cycles after starting study treatment until end of treatment; expected duration approximately 12 months
  cycle = 28 days
Progression-free survival (PFS) | Every 2 cycles after starting study treatment until disease progression; expected duration approximately 12 months
  cycle = 28 days
Overall survival (OS) - only for dose expansion | From time of start treatment until the date of death; expected duration approximately 12 months
  cycle = 28 days
Plasma concentrations of LXH254 | Cycle 1 days 1, 2, 3, 8, 15, and 16; Cycle 2 days 1 and 15; Cycle 3 Day 1; Cycle 5 Day 1
  cycle = 28 days
Derived PK parameters of LXH254: Area Under the Curve (AUC) | Cycle 1 days 1, 2, 3, 8, 15, and 16; Cycle 2 days 1 and 15; Cycle 3 Day 1; Cycle 5 Day 1
  cycle = 28 days
Derived PK parameters of LXH254: Peak Plasma Concentration (Cmax) | Cycle 1 days 1, 2, 3, 8, 15, and 16; Cycle 2 days 1 and 15; Cycle 3 Day 1; Cycle 5 Day 1
  cycle = 28 days
Derived PK parameters of LXH254: Time to Peak Plasma Concentration (Tmax) | Cycle 1 days 1, 2, 3, 8, 15, and 16; Cycle 2 days 1 and 15; Cycle 3 Day 1; Cycle 5 Day 1
  cycle = 28 days
Derived PK parameters of LXH254: half-life (T1/2) | Cycle 1 days 1, 2, 3, 8, 15, and 16; Cycle 2 days 1 and 15; Cycle 3 Day 1; Cycle 5 Day 1
  cycle = 28 days
Changes from baseline of pharmacodynamics (PD) marker DUSP6 in tumor tissue and in blood | Cycle 1 day 1, 2, 3, 15, and 16; upon disease progression (expected duration approximately 12 months)
  cycle = 28 days
Plasma concentrations of PDR001 | Cycle 1 days 1, 2, 8, and 15; Cycle 2 days 1; Cycle 3 Day 1, 2 and 8; Cycle 4 Day 1; Cycle 5 Day 1; Cycle 6 Day 1
  cycle = 28 days
Derived PK parameters of PDR001: Area Under the Curve (AUC) | Cycle 1 days 1, 2, 8, and 15; Cycle 2 days 1; Cycle 3 Day 1, 2 and 8; Cycle 4 Day 1; Cycle 5 Day 1; Cycle 6 Day 1
  cycle = 28 days
Derived PK parameters of PDR001: Peak Plasma Concentration (Cmax) | Cycle 1 days 1, 2, 8, and 15; Cycle 2 days 1; Cycle 3 Day 1, 2 and 8; Cycle 4 Day 1; Cycle 5 Day 1; Cycle 6 Day 1
  cycle = 28 days
Derived PK parameters of PDR001: Time to Peak Plasma Concentration (Tmax) | Cycle 1 days 1, 2, 8, and 15; Cycle 2 days 1; Cycle 3 Day 1, 2 and 8; Cycle 4 Day 1; Cycle 5 Day 1; Cycle 6 Day 1
  cycle = 28 days
Derived PK parameters of PDR001: half-life (T1/2) | Cycle 1 days 1, 2, 8, and 15; Cycle 2 days 1; Cycle 3 Day 1, 2 and 8; Cycle 4 Day 1; Cycle 5 Day 1; Cycle 6 Day 1
  cycle = 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (17):
- United States (3):
  - Massachusetts General Hospital MGH Cancer Center, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center SC - LXH254X2101, New York, New York
  - UT M.D Anderson Cancer Center SC - LXH254X2101, Houston, Texas
- Novartis Investigative Site, Toronto, Ontario, Canada
- France (2):
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Toulouse
- Novartis Investigative Site, Heidelberg, Germany
- Italy (3):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Napoli
- Novartis Investigative Site, Chuo Ku, Tokyo, Japan
- Netherlands (2):
  - Novartis Investigative Site, Groningen
  - Medical Oncology, Erasmus MC, Rotterdam
- Novartis Investigative Site, Seoul, South Korea
- Spain (2):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study Results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18004